CLINICAL TRIAL: NCT05905783
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter, Phase 3 Study to Evaluate the Efficacy and Safety of Izokibep in Subjects With Moderate to Severe Hidradenitis Suppurativa
Brief Title: Hidradenitis Suppurativa Study of Izokibep
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Per our 13Aug24 press release, we announced discontinuation of internal development in this indication. This decision was not due to safety reasons.
Sponsor: ACELYRIN Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 22107; 2022-503160-33-00 (Other: EU Clinical Trial Number)
Record Dates: First submitted 2023-06-07; First posted 2023-06-15 (Actual); Results first posted 2025-10-15 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2024-12

CONDITIONS: Hidradenitis Suppurativa
MeSH Terms: conditions — Hidradenitis Suppurativa

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Participants will receive placebo as a subcutaneous (SC) injection every week (QW) from Day 1 to Week 15. Participants will then receive izokibep as a SC injection QW from Week 16 to Week 51.
  Interventions: Drug: Placebo; Drug: Izokibep
- Group 2 (Experimental): Participants will receive izokibep QW from Day 1 to Week 51.
  Interventions: Drug: Izokibep

INTERVENTIONS:
Drug: Placebo — Solution for injection
  Arms: Group 1
Drug: Izokibep — Solution for injection

SUMMARY:
Izokibep is a small protein molecule that acts as a selective, potent inhibitor of interleukin 17A, to which it binds with high affinity. This study investigates izokibep in participants with active Hidradenitis Suppurativa (HS), including tumor necrosis factor-alpha inhibitor (TNFi) naïve participants, and those who had an inadequate response or intolerance to TNFi, or for whom TNFi is contraindicated.

ELIGIBILITY:
Inclusion Criteria:

General

* Participant has provided signed informed consent including consenting to comply with the requirements and restrictions listed in the informed consent form (ICF) and in protocol
* 18 years of age or older
* No known history of active tuberculosis unless adequately treated according to World Health Organization/Center for Disease Control and Prevention therapeutic guidance and determined to be fully recovered by a tuberculosis specialist

Type of Participant and Disease Characteristics

* Diagnosis of HS for ≥ 6 months prior to first dose of study drug
* Hidradenitis suppurativa lesions present in ≥ 2 distinct anatomic areas, one of which is Hurley Stage II or Hurley Stage III
* A total AN count of ≥ 5 at screening and Day 1 prior to enrollment/randomization
* Participant must have had an inadequate response to oral antibiotics OR exhibited recurrence after discontinuation to, OR demonstrated intolerance to, OR have a contraindication to oral antibiotics for treatment of their HS
* Must agree to use daily or a minimum of 3 days a week over-the-counter topical antiseptics
* Participant must be willing to complete a daily skin pain diary

Exclusion Criteria:

Medical Conditions

* Draining fistula count of > 20
* Outpatient surgery ≤ 8 weeks prior or inpatient surgery ≤ 12 weeks prior to enrollment/randomization
* Other active skin disease or condition that could interfere with study assessments
* History of active inflammatory bowel disease (IBD) OR symptoms within the last year that may be suggestive of IBD
* Chronic pain not associated with HS
* Uncontrolled, clinically significant system disease
* History of demyelinating disease or neurological symptoms suggestive of demyelinating disease
* Malignancy within 5 years
* The participant is at risk of self-harm or harm to others
* Active infection or history of certain infections
* Tuberculosis or fungal infection seen on available chest x-ray taken within 3 months prior to first dose of study drug or at screening (Exception: documented evidence of completed treatment and clinically resolved)
* Known history of human immunodeficiency virus (HIV)

Other protocol defined Inclusion/Exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Actual)
Dates: Start 2023-06-22 (Actual); Primary Completion 2024-07-24 (Actual); Study Completion 2025-01-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shephard Mpofu, Study Director — ACELYRIN Inc.
Locations (90):
- United States (47):
  - Clinical Research Site, Birmingham, Alabama
  - Clinical Research Site, Scottsdale, Arizona
  - Clinical Research Site, Fayetteville, Arkansas
  - Clinical Research Site, Encino, California
  - Clinical Research Site, Fountain Valley, California
  - Clinical Research Site, Fremont, California
  - Clinical Research Site, Los Angeles, California
  - Clinical Research Site, Santa Monica, California
  - Clinical Research Site, Boca Raton, Florida
  - Clinical Research Site, Brandon, Florida
  - Clinical Research Site, Coral Gables, Florida
  - Clinical Research Site, Hollywood, Florida
  - Clinical Research Site, Tampa, Florida
  - Clinical Research Site, Atlanta, Georgia
  - Clinical Research Site, Sandy Springs, Georgia
  - Clinical Research Site, Savannah, Georgia
  - Clinical Research Site, Springfield, Illinois
  - Clinical Research Site, Indianapolis, Indiana
  - Clinical Research Site, Plainfield, Indiana
  - Clinical Research Site, Topeka, Kansas
  - Clinical Research Site, Murray, Kentucky
  - Clinical Research Site, Baton Rouge, Louisiana
  - Clinical Research Site, New Orleans, Louisiana
  - Clinical Research Site, Largo, Maryland
  - Clinical Research Site, Boston, Massachusetts
  - Clinical Research Site, Canton, Michigan
  - Clinical Research Site, Troy, Michigan
  - Clinical Research Site, Lebanon, New Hampshire
  - Clinical Research Site, New York, New York
  - Clinical Research Site, Charlotte, North Carolina
  - Clinical Research Site, Boardman, Ohio
  - Clinical Research Site, Mason, Ohio
  - Clinical Research Site, Springfield, Ohio
  - Clinical Research Site, Portland, Oregon
  - Clinical Research Site, Hershey, Pennsylvania
  - Clinical Research Site, Pittsburgh, Pennsylvania
  - Clinical Research Site, Sugarloaf, Pennsylvania
  - Clinical Research Site, Thompson's Station, Tennessee
  - Clinical Research Site, Arlington, Texas
  - Clinical Research Site, Frisco, Texas
  - Clinical Research Site, Pflugerville, Texas
  - Clinical Research Site, San Antonio, Texas
  - Clinical Research Site, The Woodlands, Texas
  - Clinical Research Site, Webster, Texas
  - Clinical Research Site, Springville, Utah
  - Clinical Research Site, West Jordan, Utah
  - Clinical Research Site, Charlottesville, Virginia
- Canada (7):
  - Clinical Research Site, Edmonton, Alberta
  - Clinical Research Site, Winnipeg, Manitoba
  - Clinical Research Site, North Bay, Ontario
  - Clinical Research Site, Peterborough, Ontario
  - Clinical Research Site, Toronto, Ontario
  - Clinical Research Site, Waterloo, Ontario
  - Clinical Research Site, Saskatoon, Saskatchewan
- France (4):
  - Clinical Research Site, Dijon, Bourgogne-Franche-Comté
  - Clinical Research Site, Montpellier, Occitanie
  - Clinical Research Site, Nantes, Pays de la Loire Region
  - Clinical Research Site, Toulon
- Germany (5):
  - Clinical Research Site, Darmstadt, Hesse
  - Clinical Research Site, Bad Bentheim, Lower Saxony
  - Clinical Research Site, Mainz, Rhineland-Palatinate
  - Clinical Research Site, Leipzig, Saxony
  - Clinical Research Site, Kiel, Schleswig-Holstein
- Hungary (3):
  - Clinical Research Site, Debrecen, Hajdú-Bihar
  - Clinical Research Site, Zalaegerszeg, Zala County
  - Clinical Research Site, Budapest
- Japan (11):
  - Clinical Research Site, Fukuoka, Fukoka Prefecture
  - Clinical Research Site, Kitakyushu, Fukuoka
  - Clinical Research Site, Obihiro, Hokkaido Prefecture
  - Clinical Research Site, Sapporo, Hokkaido Prefecture
  - Clinical Research Site, Kawasaki, Kanagawa
  - Clinical Research Site, Yokohama, Kanagawa
  - Clinical Research Site, Kyoto, Kyoto
  - Clinical Research Site, Osaka, Osaka
  - Clinical Research Site, Shinjuku-Ku, Tokyo
  - Clinical Research Site, tabashi City, Tokyo
  - Clinical Research Site, Nishinomiya
- Poland (7):
  - Clinical Research Site, Krakow, Lesser Poland Voivodeship
  - Clinical Research Site, Wroclaw, Lower Silesian Voivodeship
  - Clinical Research Site, Lublin, Lublin Voivodeship
  - Clinical Research Site, Katowice, Silesian Voivodeship
  - Clinical Research Site, Ożarowice, Silesian Voivodeship
  - Clinical Research Site, Sosnowiec, Silesian Voivodeship
  - Clinical Research Site, Lodz, Łódź Voivodeship
- Spain (6):
  - Clinical Research Site, Seville, Andalusia
  - Clinical Research Site, Palma de Mallorca, Balearic Islands
  - Clinical Research Site, Badalona, Catalonia
  - Clinical Research Site, Barcelona, Catalonia
  - Clinical Research Site, Manises, Valencia
  - Clinical Research Site, Madrid

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 258 participants were enrolled in Canada, France, Germany, Japan, Poland, Spain and the United States from June 2023 to January 2025. Participants were randomized to receive izokibep or placebo once weekly (QW) until Week 15 (Period 1). Then, all participants received izokibep QW from Week 16 until Week 51 (Period 2).
  The Sponsor decided to terminate the study early after all participants completed (or discontinued) treatment at Week 32.
Groups:
- Placebo-Izokibep 160 mg QW: Participants received placebo as a subcutaneous (SC) injection QW from Day 1 to Week 15, then izokibep as a SC injection QW from Week 16 to Week 51.
- Izokibep 160 mg QW: Participants received izokibep as a SC injection QW from Day 1 to Week 51.
Period: Overall Study
Arm/Group | Placebo-Izokibep 160 mg QW | Izokibep 160 mg QW
Started | 129 | 129
Completed Period 1 | 109 | 103
Completed | 19 | 9
Not Completed | 110 | 120
Not completed — Lost to Follow-up | 12 | 18
Not completed — Withdrawal by Subject | 29 | 37
Not completed — Decision by sponsor | 69 | 65

BASELINE CHARACTERISTICS:
Groups:
- Placebo-Izokibep 160 mg QW: Participants received placebo as a SC injection QW from Day 1 to Week 15, then izokibep as a SC injection QW from Week 16 to Week 51.
- Izokibep 160 mg QW: Participants received izokibep QW from Day 1 to Week 51.
- Total: Total of all reporting groups
Arm/Group | Placebo-Izokibep 160 mg QW | Izokibep 160 mg QW | Total
Number analyzed (Participants) | 129 | 129 | 258
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 125 | 127 | 252
  >=65 years | 4 | 2 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.4 (12.85) | 37.1 (11.89) | 37.3 (12.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 89 | 89 | 178
  Male | 40 | 40 | 80
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18 | 12 | 30
  Not Hispanic or Latino | 108 | 115 | 223
  Unknown or Not Reported | 3 | 2 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 3 | 3
  Asian | 10 | 8 | 18
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 28 | 21 | 49
  White | 90 | 91 | 181
  More than one race | 0 | 0 | 0
  Other | 1 | 5 | 6

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Hidradenitis Suppurativa Clinical Response 75 (HiSCR75) at Week 12
Description: The percentage of participants achieving HiSCR75 was defined as meeting all 3 criteria below:
  * ([abscess and inflammatory nodule (AN) count at baseline - AN count at current visit] / AN count at baseline) × 100% ≥ 75%
  * Abscess count at baseline ≥ abscess count at the current visit
  * Draining fistula count at baseline ≥ draining fistula count at the current visit.
  HiSCR75 was evaluated using nonresponse imputation (NRI) and multiple imputation (MI) methods.
Time Frame: Week 12
Population: Full Analysis Set: all participants who were randomized.
Measure: Mean (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo-Izokibep 160 mg QW | Izokibep 160 mg QW
Number analyzed (Participants) | 129 | 129
percentage of participants | 20.3 [13.1 to 27.6] | 32.6 [24.3 to 40.9]
Statistical Analysis 1: Comparison: Placebo-Izokibep 160 mg QW vs Izokibep 160 mg QW; Test type: Superiority; p = 0.0183, Cochran-Mantel-Haenszel; Risk Difference (RD) = 13.0, 95% CI 2-sided [2.2 to 23.7], Standard Error of Mean 5.50

2. Secondary Outcome: Percentage of Participants Achieving HiSCR90 at Week 12
Description: The percentage of participants achieving HiSCR90 was defined as meeting all 3 criteria below:
  * ([AN count at baseline - AN count at current visit] / AN count at baseline) × 100% ≥ 90%
  * Abscess count at baseline ≥ abscess count at the current visit
  * Draining fistula count at baseline ≥ draining fistula count at the current visit.
  HiSCR90 was evaluated using nonresponse imputation (NRI) and multiple imputation (MI) methods.
Time Frame: Week 12
Population: Full Analysis Set: all participants who were randomized.
Measure: Mean (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo-Izokibep 160 mg QW | Izokibep 160 mg QW
Number analyzed (Participants) | 129 | 129
percentage of participants | 9.2 [3.8 to 14.5] | 24.3 [16.7 to 31.9]
Statistical Analysis 1: Comparison: Placebo-Izokibep 160 mg QW vs Izokibep 160 mg QW; Test type: Superiority; p = 0.0007, Cochran-Mantel-Haenszel; Risk Difference (RD) = 15.8, 95% CI 2-sided [6.7 to 25.0], Standard Error of Mean 4.67

3. Secondary Outcome: Percentage of Participants Achieving HiSCR100 at Week 12
Description: The percentage of participants achieving HiSCR100 was defined as meeting all 3 criteria below:
  * ([AN count at baseline - AN count at current visit] / AN count at baseline) × 100% = 100%
  * Abscess count at baseline ≥ abscess count at the current visit
  * Draining fistula count at baseline ≥ draining fistula count at the current visit.
  HiSCR100 was evaluated using nonresponse imputation (NRI) and multiple imputation (MI) methods.
Time Frame: Week 12
Population: Full Analysis Set: all participants who were randomized.
Measure: Mean (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo-Izokibep 160 mg QW | Izokibep 160 mg QW
Number analyzed (Participants) | 129 | 129
percentage of participants | 7.3 [2.5 to 12.2] | 21.4 [14.2 to 28.7]
Statistical Analysis 1: Comparison: Placebo-Izokibep 160 mg QW vs Izokibep 160 mg QW; Test type: Superiority; p = 0.0008, Cochran-Mantel-Haenszel; Risk Difference (RD) = 14.7, 95% CI 2-sided [6.1 to 23.4], Standard Error of Mean 4.40

4. Secondary Outcome: Percentage of Participants Achieving HiSCR50 at Week 12
Description: The percentage of participants achieving HiSCR50 was defined as meeting all 3 criteria below:
  * [(AN count at baseline - AN count at current visit) / AN count at baseline] × 100% ≥ 50%
  * Abscess count at baseline ≥ abscess count at the current visit
  * Draining fistula count at baseline ≥ draining fistula count at the current visit.
  HiSCR50 was evaluated using nonresponse imputation (NRI) and multiple imputation (MI) methods.
Time Frame: Week 12
Population: Full Analysis Set: all participants who were randomized.
Measure: Mean (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo-Izokibep 160 mg QW | Izokibep 160 mg QW
Number analyzed (Participants) | 129 | 129
percentage of participants | 36.5 [27.8 to 45.2] | 47.9 [39.0 to 56.8]
Statistical Analysis 1: Comparison: Placebo-Izokibep 160 mg QW vs Izokibep 160 mg QW; Test type: Superiority; p = 0.0462, Cochran-Mantel-Haenszel; Risk Difference (RD) = 12.3, 95% CI 2-sided [0.2 to 24.3], Standard Error of Mean 6.16

5. Secondary Outcome: Percentage of Participants Who Experienced One or More (≥ 1) Disease Flare at Week 12
Description: HS flares were defined as ≥ 25% increase in AN count with a minimum increase of 2 AN relative to baseline, i.e. participants must meet all the following criteria:
  * (AN count at current visit- AN count at baseline) / AN count at baseline ×100% ≥ 25%
  * AN count at current visit- AN count at baseline ≥ 2.
  Participants who received antibiotic therapy that could affect HS were imputed as non-response (NRI). Other participants with missing data were imputed with multiple imputation.
Time Frame: Up to Week 12
Population: Full Analysis Set: all participants who were randomized.
Measure: Mean (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo-Izokibep 160 mg QW | Izokibep 160 mg QW
Number analyzed (Participants) | 129 | 129
percentage of participants | 31.1 [22.9 to 39.3] | 28.3 [20.5 to 36.2]
Statistical Analysis 1: Comparison: Placebo-Izokibep 160 mg QW vs Izokibep 160 mg QW; Test type: Superiority; p = 0.6285, Cochran-Mantel-Haenszel; Risk Difference (RD) = -2.8, 95% CI 2-sided [-14.3 to 8.6], Standard Error of Mean 5.84

6. Secondary Outcome: Change From Baseline in Dermatology Life Quality Index (DLQI)
Description: DLQI included 10 items arranged in 6 categories: symptoms and feelings, daily activity, leisure, work or study, interpersonal relationships, and treatment. The total score could range from 0 (no impact to life quality) to 30 (maximum impact).
Time Frame: Baseline and Week 12
Population: Full Analysis Set: all participants who were randomized. Only participants with a result at the timepoint are included.
Measure: Least Squares Mean (Standard Error); unit: Score on scale
Arm/Group | Placebo-Izokibep 160 mg QW | Izokibep 160 mg QW
Number analyzed (Participants) | 112 | 102
Score on scale | -2.71 (0.519) | -4.87 (0.536)
Statistical Analysis 1: Comparison: Placebo-Izokibep 160 mg QW vs Izokibep 160 mg QW; Test type: Superiority; p = 0.0011, Mixed model repeated measures (MMRM); LS Mean Difference = -2.16, 95% CI 2-sided [-3.44 to -0.88]

7. Secondary Outcome: Percentage of Participants With Baseline Hurley Stage II Who Achieved AN Count of 0, 1, or 2 at Week 12
Description: Calculated as observed values of 0, 1, or 2 for AN count (abscess count + inflammatory nodule count).
  AN count of 0, 1, or 2 was evaluated using nonresponse imputation (NRI) and multiple imputation (MI) methods.
Time Frame: Week 12
Population: Full Analysis Set: all participants who were randomized. Participants with Hurley Stage II at baseline were included.
Measure: Mean (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo-Izokibep 160 mg QW | Izokibep 160 mg QW
Number analyzed (Participants) | 82 | 78
percentage of participants | 25.0 [15.2 to 34.8] | 49.5 [38.1 to 61.0]
Statistical Analysis 1: Comparison: Placebo-Izokibep 160 mg QW vs Izokibep 160 mg QW; Test type: Superiority; p = 0.0013, Cochran-Mantel-Haenszel; Risk Difference (RD) = 24.6, 95% CI 2-sided [9.6 to 39.7], Standard Error of Mean 7.67

8. Secondary Outcome: Percentage of Participants With Baseline NRS ≥ 4 Achieving at Least 3-point Reduction at Week 12 in Numeric Rating Scale (NRS) Patient Global Assessment of Skin Pain at Its Worst
Description: NRS in Patient Global Assessment of Skin Pain ranged from 0 (no skin pain) to 10 (skin pain bad as you can imagine). The skin pain score at each visit was calculated using average of daily scores among the 7 days up to and including the day of visit, with a minimum of 4 days (consecutive or non-consecutive) with scores required.
  Reduction in NRS was evaluated using nonresponse imputation (NRI) and multiple imputation (MI) methods.
Time Frame: Week 12
Population: Full Analysis Set: all participants who were randomized. Participants with baseline NRS ≥ 4 were included.
Measure: Mean (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo-Izokibep 160 mg QW | Izokibep 160 mg QW
Number analyzed (Participants) | 79 | 73
Percentage of participants | 17.2 [8.4 to 25.9] | 33.5 [22.1 to 44.8]
Statistical Analysis 1: Comparison: Placebo-Izokibep 160 mg QW vs Izokibep 160 mg QW; Test type: Superiority; p = 0.0245, Cochran-Mantel-Haenszel; Risk Difference (RD) = 16.3, 95% CI 2-sided [2.1 to 30.6], Standard Error of Mean 7.26

9. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs), Serious AEs (SAEs) and Adverse Event of Special Interest (AESIs) in Period 1
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study drug, whether or not considered related to the study drug.
  An SAE is defined as any untoward medical occurrence that, at any dose, meets one or more of the criteria listed: results in death, is life threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, or is an important medical event.
  The following events of special interest were monitored in this study: candida infection; inflammatory bowel disease (IBD); suicidal ideation; malignancies; major adverse cardiovascular and cerebrovascular events; tuberculosis; infections; cytopenias and systemic hypersensitivity reactions.
  Clinically significant changes in vital signs and laboratory tests recorded after treatment administration were documented as TEAEs.
Time Frame: Up to Week 16
Population: Safety Analysis Set: All participants who were randomized and received at least 1 administration of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo-Izokibep 160 mg QW | Izokibep 160 mg QW
Number analyzed (Participants) | 129 | 129
Participants
  TEAEs | 76 | 107
  SAEs | 5 | 1
  AESIs | 3 | 0

10. Secondary Outcome: Number of Participants With TEAEs, SAEs and AESIs in Period 2
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study drug, whether or not considered related to the study drug.
  An SAE is defined as any untoward medical occurrence that, at any dose, meets one or more of the criteria listed: results in death, is life threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, or is an important medical event.
  The following events of special interest were monitored in this study: candida infection; IBD; suicidal ideation; malignancies; major adverse cardiovascular and cerebrovascular events; tuberculosis; infections; cytopenias and systemic hypersensitivity reactions.
  Clinically significant changes in vital signs and laboratory tests recorded after treatment administration were documented as TEAEs.
Time Frame: From Week 16 to follow-up, Week 59
Population: Safety Analysis Set Period 2: All participants who were randomized and received at least 1 administration of study treatment in Period 2 of the Study.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo-Izokibep 160 mg QW | Izokibep 160 mg QW
Number analyzed (Participants) | 109 | 100
Participants
  TEAEs | 87 | 66
  SAEs | 3 | 4
  AESIs | 5 | 1

ADVERSE EVENTS:
Time Frame: From Screening (Day -28) to Follow-up (Week 59), up to approximately 63 weeks
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study drug, whether or not considered related to the study drug.
  Safety Analysis Set: All participants who were randomized and received at least 1 administration of study treatment.
Groups:
- Placebo QW - Izokibep 160 mg QW: Period 1: Participants received placebo as a SC injection QW from Day 1 to Week 15.
- Izokibep 160 mg QW: Period 1: Participants received izokibep QW from Day 1 to Week 15.
- Placebo QW - Izokibep 160 mg QW: Period 2: Participants received izokibep as a SC injection QW from Week 16 to Week 51.
- Izokibep 160 mg QW: Period 2: Participants received izokibep QW from Week 16 to Week 51.
Arm/Group | Placebo QW - Izokibep 160 mg QW: Period 1 | Izokibep 160 mg QW: Period 1 | Placebo QW - Izokibep 160 mg QW: Period 2 | Izokibep 160 mg QW: Period 2
All-Cause Mortality (participants affected / at risk) | 0/129 | 0/129 | 0/109 | 0/100
Serious Adverse Events (participants affected / at risk) | 5/129 | 1/129 | 3/109 | 4/100
Other Adverse Events (participants affected / at risk) | 35/129 | 93/129 | 69/109 | 40/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo QW - Izokibep 160 mg QW: Period 1 (N=129) | Izokibep 160 mg QW: Period 1 (N=129) | Placebo QW - Izokibep 160 mg QW: Period 2 (N=109) | Izokibep 160 mg QW: Period 2 (N=100)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hidradenitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Vasculitis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye disorder (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo QW - Izokibep 160 mg QW: Period 1 (N=129) | Izokibep 160 mg QW: Period 1 (N=129) | Placebo QW - Izokibep 160 mg QW: Period 2 (N=109) | Izokibep 160 mg QW: Period 2 (N=100)
Injection site reaction (General disorders) | 10 (16) | 86 (380) | 66 (328) | 34 (186)
Fatigue (General disorders) | 3 (3) | 7 (12) | 0 (0) | 2 (2)
Nasopharyngitis (Infections and infestations) | 9 (12) | 11 (11) | 5 (5) | 8 (9)
Upper respiratory tract infection (Infections and infestations) | 5 (6) | 7 (7) | 5 (5) | 4 (5)
Headache (Nervous system disorders) | 16 (37) | 14 (26) | 2 (2) | 5 (6)
Diarrhoea (Gastrointestinal disorders) | 2 (3) | 7 (7) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2024-05-14): https://cdn.clinicaltrials.gov/large-docs/83/NCT05905783/Prot_000.pdf
  • Statistical Analysis Plan (2024-12-10): https://cdn.clinicaltrials.gov/large-docs/83/NCT05905783/SAP_001.pdf